CLINICAL TRIAL: NCT04238754
Title: A Randomized Placebo-Controlled Evaluation of the Safety of Oral Cannabidiol in a Clinically Relevant Model of Opioid Withdrawal
Brief Title: Oral Cannabidiol for Opioid Withdrawal
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Dalio Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00232412
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Opioid Withdrawal; Opioid Craving; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Within subject comparison of Epidiolex to placebo. The order of study drug (active Epidiolex or placebo) is randomized across participants. Epidiolex is flavor masked with cherry syrup.
Masking Description: Epidiolex is flavor masked with cherry syrup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epidiolex (CBD) Then Placebo (Experimental): Participants first receive 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses) during which prescribed methadone is withheld. After 1 week, they receive 20 mL of inactive cherry syrup delivered every 12 hours for 48hours total (4 doses) during which prescribed methadone is withheld.
  Interventions: Drug: Epidiolex; Drug: Placebo
- Placebo Then Epidiolex (Placebo Comparator): Participants first receive 20 mL of inactive cherry syrup delivered every 12 hours for 48hours total (4 doses) during which prescribed methadone is withheld. After 1 week washout, they receive 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses) during which prescribed methadone is withheld.
  Interventions: Drug: Epidiolex; Drug: Placebo

INTERVENTIONS:
Drug: Epidiolex — Epidiolex 100 mg/mL Oral Solution
  Other Names: Cannabidiol
Drug: Placebo — Cherry syrup oral solution

SUMMARY:
This pilot study will examine the safety of the cannabinoid cannabidiol (Epidiolex) in a human laboratory model of clinically relevant withdrawal. The study will be a residential within-subject comparison; all participants will receive placebo dosing and active cannabidiol. Results may be used to support an R01 grant application to more closely examine this hypothesis.

DETAILED DESCRIPTION:
Based on preclinical research and emerging human research, cannabidiol (CBD; a major constituent of the cannabis plant) is a promising pharmacotherapy for the treatment of opioid withdrawal. Most recently, CBD decreased cue-induced craving and anxiety (two common withdrawal symptoms) among abstinent heroin-dependent individuals relative to placebo. As of June 2018, Epidiolex, an oral formulation of plant-derived pure CBD, has been approved by the U.S. Food and Drug Administration (FDA) for treating severe forms of epilepsy and can be prescribed for other off-label indications. Epidiolex has a low side effect and high safety profile. Given the recent FDA approval of Epidiolex, and a growing interest to develop existing pharmaceuticals to address issues related to Opioid Use Disorder (OUD) and its recovery, the investigators are proposing a pilot study to examine the safety of Epidiolex in a human laboratory model of clinically relevant withdrawal. The study will be a residential within-subject comparison; methadone-maintained participants will undergo spontaneous withdrawal and receive placebo dosing and active cannabidiol. Data collected for this study will establish: (1) the safety of administering two dosing regimens of Epidiolex within the investigators' withdrawal paradigm and (2) the feasibility of the investigators' withdrawal paradigm for demonstrating clinically meaningful increases in withdrawal. Results may be used to support an R01 grant application to more closely examine this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Medically cleared to take study medication
* Are not pregnant or breast feeding
* Willing to comply with the study protocol
* Provides urine that tests positive for methadone
* Maintained on 80-120 mg of daily methadone with no dose changes in the past 2 weeks (verified through a medical release with the participant's provider)

Exclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for alcohol/substance use disorder other than opioid use disorder
* Previous adverse reaction to a cannabinoid product
* Self-report any illicit drug use or cannabinoid use in the past 7 days
* Presence of any clinically significant medical/psychiatric illness judged by the investigators to put subject at elevated risk for experiencing an adverse events
* Past year suicidal behavior as assessed via the Columbia Suicide Severity Rating Scale
* History of seizure disorder
* Past 14 day use of any of the following contraindicated medications:

  * Clobazam, Valproate
  * Moderate or strong inhibitors of CYP3A4 or CYPC19 (with the exception of methadone, as outlined in the Protection Against CBD Risks section).
  * Strong CYP3A4 or CYP2C19 inducers
  * UGT1A9, UGT2B7, CYP1A2, CYP2C8, CYP2C9 and CYP2C19 substrates (with the exclusion of caffeine).
  * Central nervous system (CNS) depressants that are contraindicated with Epidiolex
* Breathalyzer that tests positive for alcohol prior to session admission
* Self-reported consumption of grapefruit juice within 24 hours of session admission
* Have a history of clinically significant cardiac arrhythmias or vasospastic disease
* Have circumstances that the study investigators believe are contraindicated with study participation and/or would interfere with study participation (e.g., impending jail).
* Moderate-severe hepatic impairment as indicated by ALT or AST levels > 3x ULN and/or Bilirubin levels >2x ULN as evidenced by a blood test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia L Bergeria, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidiolex Then Placebo: Participants first receive 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses) during which prescribed methadone is withheld. After 1 week, they receive 20 mL of inactive cherry syrup delivered every 12 hours for 48hours total (4 doses) during which prescribed methadone is withheld.
Period: First Intervention
Arm/Group | Epidiolex Then Placebo | Placebo Then Epidiolex
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Washout - 1 Week
Arm/Group | Epidiolex Then Placebo | Placebo Then Epidiolex
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention
Arm/Group | Epidiolex Then Placebo | Placebo Then Epidiolex
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each participant will receive Epidiolex oral solution and Cherry syrup oral solution (placebo) in a randomized fashion.
  Epidiolex 100 mg/mL Oral Solution: 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
  Cherry Syrup Oral Solution: 20 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Number of Adverse Events
Description: Number of Adverse Events reported across sessions with and without study drug. Adverse events were collected for the entire 57 hour session.
Time Frame: through completion of the two study sessions, an average of 17 days
Measure: Number; unit: Adverse Events
Arm/Group | All Participants
Number analyzed (Participants) | 3
Adverse Events
  Placebo Adverse Events | 4
  Epidiolex Adverse Events | 5

2. Primary Outcome: Number of Participants Whose Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) Levels >3x Upper Limit of Normal
Description: Number of participants whose AST/ALT levels >3x upper limit of normal (ULN) at the end of a study session when they receive Epidiolex and Placebo. This will be used in the assessment of safety.
Time Frame: End of residential stay, prior to discharge
Measure: Count of Participants; unit: Participants
Groups:
- Epidiolex; Placebo: Each participant will receive Epidiolex oral solution and Cherry syrup oral solution (placebo) in a randomized fashion.
  Epidiolex 100 mg/mL Oral Solution: 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
  Cherry Syrup Oral Solution: 20 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
Arm/Group | Epidiolex | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

3. Primary Outcome: Change in Withdrawal Scores From Baseline AfterReceiving Placebo
Description: Change in withdrawal scores during laboratory evaluation of spontaneous withdrawal. Withdrawal is measured with the Subjective Opiate Withdrawal Scale (SOWS). That has a range of 0-64 where a mild score is represented by a score of 1-10, a moderate score is represented by a score of 11-20 and a severe score is considered anything greater than 21.
Time Frame: Baseline, during residential session up to 57 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 3
score on a scale | 15.8 (6.3)

4. Secondary Outcome: Initial Efficacy of Study Drug as Assessed by Area Under the Curve for the Subjective Opiate Withdrawal Scale (SOWS) Scores
Description: Withdrawal symptom suppression during active and placebo conditions. Area Under the Curve (AUC) analyses will be calculated to characterize withdrawal on the Subjective Opiate Withdrawal Scale (SOWS) scores across time. SOWS AUC will be compared between the two conditions. AUC will range from 0 to 3072 where 0 represents no withdrawal during study drug administration and 3072 represents the most severe withdrawal during study drug administration.
Time Frame: After first administration of study drug and up to 48 hours
Measure: Mean (Standard Deviation); unit: scores on SOWS scale X hour
Groups:
- Placebo: Flavor-matched placebo syrup
Arm/Group | Epidiolex | Placebo
Number analyzed (Participants) | 3 | 2
scores on SOWS scale X hour | 1334.7 (57.8) | 1591.5 (12.0)

5. Secondary Outcome: Acceptability Assessed by Number of Participants Who Would Recommend the Medication to a Family Member or Friend
Description: Number of participants who would recommend the medication to a family member or friend trying to taper down from opioid medications.
Time Frame: at the end of the 57-hour residential session, prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Epidiolex | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

6. Secondary Outcome: Acceptability Assessed by Visual Analog Ratings
Description: Visual analog ratings of the degree to which the medication suppressed opioid withdrawal symptoms. The visual analog ratings will be scored on a scale from 0-100 where 0 represents no suppression of withdrawal and 100 represents complete suppression of withdrawal.
Time Frame: at the end of the 57-hour residential session, prior to discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidiolex | Placebo
Number analyzed (Participants) | 3 | 2
units on a scale | 24.333 (9.0) | 17.5 (3.5)

7. Secondary Outcome: Acceptability Assessed by Rating of Medication Acceptance on a 5-point Acceptance Rating Scale
Description: Participant rating of medication acceptance on a 5-point acceptance rating scale. The acceptance rating scale will range from 0-4 where 0 represents no acceptance of the medication and 4 represents complete acceptance of the medication.
Time Frame: at the end of the 57-hour residential session, prior to discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epidiolex | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 4 (0) | 4 (0)

ADVERSE EVENTS:
Time Frame: through completion of the two study sessions, an average of 17 days
Groups:
- Epidiolex: Epidiolex 100 mg/mL oral solution: 8 mL of Epidiolex (800 mg of cannabidiol) + 16 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
- Placebo: Cherry Syrup Oral Solution: 20 mL of inactive cherry syrup delivered every 12 hours for 48 hours total (4 doses)
Arm/Group | Epidiolex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidiolex (N=3) | Placebo (N=3)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04238754/Prot_SAP_000.pdf